CLINICAL TRIAL: NCT04712266
Title: A Randomized, Double-blinded Trial to Investigate Glycemic Excursions Following an Oral Mixed Meal Challenge in Subjects With Type 1 Diabetes When Concomitantly Treated With Insulin Alone or Co-administered Insulin and Glucagon
Brief Title: A Trial to Investigate Hyperglycemic and Hypoglycemic Excursions in Subjects With Type 1 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abvance Therapeutics (Industry)
Collaborators: T1D Exchange, United States (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABV201
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia
MeSH Terms: interventions — Glucagon; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin IV (Active Comparator): calculated insulin rate
  Interventions: Drug: Insulin
- Insulin and Glucagon IV (Experimental): calculated molar ratio insulin:glucagon
  Interventions: Drug: Glucagon; Drug: Insulin

INTERVENTIONS:
Drug: Glucagon — calculated IV insulin:Glucagon molar ratio
  Other Names: Glucagen Hypokit
  Arms: Insulin and Glucagon IV
Drug: Insulin — calculated IV Insulin dose infused at a constant rate
  Other Names: Human Insulin (Eli Lilly)

SUMMARY:
This is a single center, double-blind, randomized trial in subjects with type 1 diabetes mellitus applying an adaptive design approach.

DETAILED DESCRIPTION:
Subjects were be studied on two occasions, in randomized sequence, whereby glycemic excursions are assessed following an oral mixed meal challenge while treated with either insulin alone or co-administered insulin and glucagon.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 64 years (both inclusive)
* Type 1 diabetes mellitus (as diagnosed clinically) ≥ 12 months prior to the screening visit
* Treated with daily insulin for T1DM ≥ 12 months prior to the screening visit

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
hypoglycemic excursions | 180-360 minutes post meal
  < 50mg/dl
hyperglycemic excursions | 60-120 minutes post meal
  >150mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Bode, MD, Principal Investigator — Atlanta Diabetes Associates
Locations (1):
- Atlanta Diabetes Associates, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No